CLINICAL TRIAL: NCT04122144
Title: Enhanced Viral Load Counseling and Standardized Peer Mother Support Study (ENHANCED-SPS)
Brief Title: Optimizing HIV Virologic Outcomes for Pregnant Women in Uganda
Acronym: ENHANCED-SPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Collaborators: Infectious Diseases Research Collaboration, Uganda (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REC REF 2018-074; HS 2648 (Other: Uganda national council of science and technology)
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: HIV
Keywords: pregnant woman

STUDY DESIGN:
Intervention Model Description: Comparative effectiveness cluster-randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): ENHANCED-SPS intervention implemented
  Interventions: Behavioral: ENHANCED -SPS intervention
- Control (No Intervention): Standard of care maintained. These are procedures conducted during the routine HIV care visits at the health facilities include ART card documentation as required, general/routine counseling, and adherence counseling to the non suppressors, ART drug supply based on the clinicians prescription and laboratory monitoring.

INTERVENTIONS:
Behavioral: ENHANCED -SPS intervention — a) Enhanced VL counseling: Explanation of VL & Importance of VL suppression,assessment of adherence, counseling based on VL result and schedule for next VL testing and the role of VL and the MTCT risk; b).Standardized peer mother support: includes training of peer mothers on mandatory enhanced VL counseling during the routine peer counseling and education, follow up of mothers and continued adherence counseling and disclosure support and bi-weekly phone calls to mothers to provide VL counseling and follow up
  Arms: Intervention

SUMMARY:
The ENHANCED -SPS study is a before and after cluster randomized trial that will be conducted in 14 public health facilities providing HIV care in Southwestern Uganda. The study will evaluate the effectiveness of a multi-component intervention package that targets barriers to achieving optimal viral suppression among pregnant and postpartum women infected with HIV. This will be in two phases; In Phase 1 ("Before"), all 14 clinics will have a baseline assessment of standard of care VL procedures and assess the barriers and facilitators to viral suppression for a period of 3 months. In Phase 2 ("After"), 7 clinics randomized to control arm will continue to experience standard of care counseling procedures, and 7 clinics randomized to intervention will initiate the ENHANCE-PS intervention. The Phase 2 ("After") phase I will last at least 12 months.

DETAILED DESCRIPTION:
The Investigators will test the hypothesis that the Enhanced viral load (VL) counseling and standardized peer mother support (ENHANCED-SPS) intervention will increase viral load suppression among HIV-infected pregnant and post-partum women and increase retention of mothers in care hence resulting in reduced risk of vertical transmission in south western Uganda.

Specific objectives are as follows:

1) To evaluate the effectiveness of an enhanced VL counseling and standardized peer mother support intervention on viral suppression among HIV infected pregnant women at 12 months of follow up; 2) To evaluate the effect of the enhanced counseling and peer support intervention on retention in care at 18 months postpartum follow up; The investigators will randomize 14 HIV clinics to the ENHANCED-SPS multi-component intervention vs. standard of care procedures (intervention=7 clinics and control=7 clinics,n=70 mothers/health facility) ;3) To assess the facilitators and barriers of VL and enhanced VL counseling and peer mother support intervention at 9 & 18 months of follow up.This will consider both patient and providers perspectives of the intervention implementation

ELIGIBILITY:
Inclusion Criteria:

1. All Pregnant women and breastfeeding mothers enrolled in the mother baby care points/HIV clinics with documented HIV infection
2. . HIV infected Pregnant women reporting for their first ANC within the study clinics or newly identified HIV positive mothers from the ANC clinics/breastfeeding

   Exclusion Criteria:
3. . All women who will be critically ill and unable to communicate
4. . Those not willing to consent to participate in the study
5. . Women who will not be able to understand all information concerning the study

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 980 (Estimated)
Dates: Start 2019-09-19 (Actual); Primary Completion 2021-09-19 (Estimated); Study Completion 2022-09-19 (Estimated)

PRIMARY OUTCOMES:
Viral suppression | 1 year
  The proportion of women with HIV-1 RNA suppression at 12 months of follow up to assess the effect of the intervention
Retention in care | 18 months
  The proportion of women still in care at at 12 and 18 months postpartum

SECONDARY OUTCOMES:
Mother to child transmission rate | 18 months
  The proportion of HIV free children born to the HIV positive mothers enrolled in the study at 18 months of follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Kabami, MPH, Principal Investigator — Makerere University; Moses Kamya, PhD, Principal Investigator — Makerere University; Phillipa Musoke, PhD, Principal Investigator — Makerere University
Locations (1):
- Jane Kabami, Kampala, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No